CLINICAL TRIAL: NCT07339891
Title: Experience of Staying in Intensive Care and Impact on Quality of Life
Acronym: Expe-Rea
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9771
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Stay in intensive care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It now seems well established that post-traumatic stress disorder following a stay in intensive care is one of the factors that affects patients' quality of life after they leave hospital.

Several qualitative and quantitative studies suggest that there are several factors associated with the onset of this post-traumatic stress disorder, including the absence of memory of the stay in intensive care. With this in mind, some intensive care units (in France and abroad) are implementing measures to improve the patient experience during their stay, particularly to compensate for this lack of memory: several studies show a link between the introduction of intensive care unit logbooks and a decrease in the incidence of post-traumatic stress disorder after returning home.

The aim of this research project is to measure the experience of the stay in intensive care and its possible impact on quality of life. It is therefore part of a process of implementing measures within general and cardiovascular surgical intensive care units, aimed at better assessing and improving the quality of life of patients after a stay in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Stay in intensive care > 48 hours

Exclusion Criteria:

* Admission to intensive care following scheduled surgery.
* Readmission to intensive care (previous admission within the 30 days prior).
* Patient under legal guardianship
* Inability to complete a questionnaire
* Poor reading and/or speaking comprehension of French
* Patient under guardianship or conservatorship.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patient (≥ 18 years) having a stay in intensive care > 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
ICE questionnaire score | Between 1 and 3 days after discharge from the intensive care unit.
  ICE (Impact Confidence Experience) questionnaire score:
  The scores for each letter (I, C, E) are added together or averaged.
  The higher the score, the better. This indicates a positive experience, trust, and a significant impact.
  Simple example:
  * Impact = 8/10 → The service was very helpful.
  * Trust = 9/10 → I trust this team.
  * Experience = 7/10 → My experience was quite good.
  Average ICE score = (8 + 9 + 7) ÷ 3 = 8/10
Quality of life questionnaire score (SF36) | Day 30 after discharge from hospital
  The SF-36 is a health questionnaire consisting of 36 questions.
  Each dimension receives a score from 0 to 100:
  * 100 = very good quality of life
  * 0 = very poor quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France